CLINICAL TRIAL: NCT03239899
Title: PD-1 Inhibition to Determine CNS Reservoir of HIV-Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170145; 17-N-0145
Record Dates: First submitted 2017-08-03; First posted 2017-08-04 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2023-02-13

CONDITIONS: HIV Infections
Keywords: HIV; Brain; Immunotherapy
MeSH Terms: conditions — HIV Infections | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HIV Participants (Experimental): Participants who received 200 mg of Pembrolizumab administered as a one-time intravenous infusion over 30 minutes during the treatment phase of the study.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Participants will receive one dose of 2mg/kg of pembrolizumab IV at Week 0.

SUMMARY:
Background:

HIV affects millions of people. The disease may "hide" in the brain, even in people with well-controlled HIV without cancer. Then it may "wake up" and continue. The drug pembrolizumab uses the body's immune system to fight cells like cancer cells. It is approved to treat some cancers but not HIV. Researchers want to see if it is safe for HIV-positive people without cancer. This study is not for HIV treatment; only one dose of the drug will be used.

Objective:

To learn if the drug pembrolizumab, used to treat certain cancers, is safe for HIV-positive people.

Eligibility:

Adults ages 18 and older with HIV who are in another NIH protocol

Design:

Participants will be screened with:

* Medical history
* Physical and neurological exams
* Blood tests
* Lumbar puncture. The lower back will be numbed. A needle will remove fluid from between back bones.
* FDG-PET/CT. A radioactive sugar will be injected in a thin plastic tube (catheter) inserted in an arm vein. Participants will rest for an hour, urinate, then lie in the scanner. A mask will hold the head still.
* Leukapheresis. An optional procedure at baseline. White blood cells are removed from you using a serum cell separator machine

Women who can become pregnant cannot take pembrolizumab. Men who take it must use 2 kinds of contraception.

Participants will have up to 7 more visits, which repeat some screening tests.

At 1 visit, participants will get one dose of pembrolizumab by catheter for 30 minutes. They will get allergy and pain medicines.

At 2 visits, participants will have a brain MRI. They will get a contrast agent by catheter. They will lie in a metal cylinder that takes pictures for 1-2 hours. They will get earplugs for loud sounds.

DETAILED DESCRIPTION:
Objective

In this Phase I, proof-of-concept study, we aim to determine the safety and tolerability of pembrolizumab, an FDA-approved monoclonal antibody against programmed cell death protein (PD)-1, in viremically suppressed human immunodeficiency virus-1 (HIV) positive patients. We are examining the correlation of immune activation and suppression markers in viremically suppressed HIV positive patients with the effects of pembrolizumab on immune restoration function (e.g. CD4 count, HIV viral load) and immune activation (e.g. HIV-specific T-cell responses).

Study Population

HIV is estimated to infect 37.6 million people globally, with 690,000 deaths and 1.5 million new infections occurring yearly. There is no cure. Opportunistic infections and neoplasms contribute to a large portion of mortality and morbidity within the HIV-positive population. Even in well- controlled, viremically suppressed patients, neurologic complications including HIV-associated neurocognitive disorder, continue to contribute to disease morbidity and mortality.

There is evidence that HIV reservoirs contribute to the inability to cure HIV infection. In the brain, macrophages and astrocytes harbor HIV. It is theorized that the brain is a potential reservoir for replication competent HIV. PD-1 expression is elevated in patients with HIV compared to uninfected controls. Upregulated PD-1 expression is associated with higher viral load and increased mortality in infections.1 PD-1 co-expression on regulatory T-cells has been shown to correlate with disease progression in perinatally-infected HIV-positive children. Drugs targeting the PD-1 pathway in HIV infection have shown upregulation of T-cell responses that are potentially critical to eradication of infection. Pembrolizumab is an attractive option due to its mechanism of action, although it has been rarely used in the HIV population.

Design

In this single-center, single-arm, open label, baseline-versus-treatment phase I clinical trial, twelve patients with HIV-1 infection receive a one-time dose of 200mg pembrolizumab with a baseline study period of 3 weeks, a one-day treatment phase, and a 6-month post treatment phase. Outcome measures are collected every 3 to 6 weeks for the duration of the study.

Outcome Measures

The primary outcome is the safety and tolerability of pembrolizumab, which is measured by clinical exam, laboratory studies and adverse event tabulations using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

In addition, viral and immunologic outcome measures investigating the impact of pembrolizumab on HIV-1 biology and its effects on immune function is measured in the CSF and periphery, including single copy HIV analysis, CD4+ T-cell count, PD-1 lymphocyte expression and T-cell phenotype analysis, T-cell proliferation against HIV-proteins, CSF cytokine analysis and/or CSF antibody profiling (LIPS). These additional studies offer indirect proof of a HIV viral reservoir in the CNS as well as potential efficacy of pembrolizumab in reversing immune exhaustion against latent HIV

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18 years or older
* Diagnosis of HIV-1 infection, with positive HIV 1 antibody testing
* HIV RNA less than or equal to 40 copies/mL in plasma in the last 12 or greater months
* CD4 count above 350 cells/uL
* Antiretroviral therapy for 12 months prior to trial
* Fully vaccinated against SARS-CoV-2. Fully vaccinated is defined as:

  * Two weeks out from the second dose of a two-dose vaccine series (Moderna, Pfizer-BioNTech); or
  * Two weeks out from a single-dose vaccine (Johnson & Johnson/Janssen)
* Patient must be willing and able to comply with all the aspects of trial design and follow-up.
* Patients must be able to provide informed consent
* Women of childbearing potential must agree to use contraception (defined as two forms of effective birth control), from the time of enrollment until 4 months after the last exposure to pembrolizumab
* Participants who are physically able to father a child must agree to use 2 effective methods of contraception (birth control) from the time you enroll in the study until 4 months after your last exposure to pembrolizumab

  * Effective methods of contraception for this study include:

    * hormonal contraception (birth control pills, birth control patches, injected hormones, hormonal implants or vaginal ring),
    * Intrauterine device,
    * Barrier methods (condom or diaphragm) combined with spermicide, and
    * Surgical sterilization (hysterectomy, tubal ligation, or vasectomy).
    * If you have had a hysterectomy, tubal ligation, or vasectomy (or have a partner with a hysterectomy, tubal ligation or vasectomy), you do not have to use 2 methods of birth control.

EXCLUSION CRITERIA:

* Clinically significant medical disorders that might expose the patient to undue risk of harm confound study outcomes or prevent the patient from completing the study as identified on screening studies and by patient history. Examples of such conditions include known cardiac disease such as congestive heart failure, chronic obstructive pulmonary disease, uncontrolled hypertension, kidney disease, liver disease, endocrine disease, pulmonary disease, heart disease, progressive CNS disease such as Parkinson s disease, dementia, prior tuberculosis infection or ongoing CNS opportunistic infection.
* Patient has received immunomodulatory/immunosuppressive therapy (including IV steroids but excluding local injections) in the preceding 6 months.
* Patient with known autoimmunity that would include but is not limited to disorders such as hypo/hyperthyroidism, myasthenia gravis, diabetes mellitus type 1, hemolytic anemia, and immune mediated hepatitis (but excluding patients with hypothyroidism already on thyroid replacement therapy).
* Prior history of cancer (excluding non-invasive squamous and basal cell carcinoma)
* Any opportunistic infection in the prior 2 years (excluding thrush) including latent TB (or a positive TB Quantiferon Gold test)
* Patient has received other investigational drugs within 3 months before enrollment
* Positive serological or PCR evidence of active or prior infection with HTLV-1/II, Hepatitis B or C. Patients with hepatitis B core (+), surface antibody (+), surface antigen ( ) and hepatitis B DNA (-) eligible to participate in the study (provided they are on tenofovir, lamivudine or TAF). Participants with prior hepatitis C who are hepatitis C antibody (+) but hepatitis C RNA (-) with normal liver enzymes and no evidence of cirrhosis on clinical liver ultrasound are eligible to participate in the study.
* Metal in the body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or history of welding or metal worker
* Claustrophobia
* Inability to lie comfortably on the back for up to two hours.
* Abnormal anti-thyroid panel (anti-TPO and anti-TG) test at screening visit.
* Abnormal screening/baseline blood tests exceeding any of the limits defined below or as deemed exclusionary by the investigators on review:

  * AST and ALT values >1.1 times ULN
  * Fasting triglyceride > 300 mg/dL
  * Total bilirubin >1.1 times ULN (unless participant is taking atazanavir or has Gilbert syndrome)
  * Creatinine Clearance or eGFR <60 ml/minute (adjusted for race)
  * Hemoglobin < 10 g/dL
  * Absolute neutrophil count < 1000/microliter
  * Platelet count <130,000/mm(3) (if platelet clumping is present on hematology slide review, platelet count <100,000/mm3 is considered exclusionary to study)
  * Hemoglobin A1c greater than or equal to 6%
  * Thyroid-stimulating hormone (TSH) and adrenocorticotropic hormone (ACTH) within normal limits. If TSH is not within normal limits then the participant may be eligible if thyroxine (T4) is within normal limits. Participants are not excluded if they are on a stable dose of replacement thyroid medication; dose may be adjusted as needed.
* An employee or staff of the NIH

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication, or at the time of publication
Access Criteria: At request, through existing NIH technology transfer policy methods

REFERENCES:
- [Derived] Henderson LJ, Reoma LB, Kovacs JA, Nath A. Advances toward Curing HIV-1 Infection in Tissue Reservoirs. J Virol. 2020 Jan 17;94(3):e00375-19. doi: 10.1128/JVI.00375-19. Print 2020 Jan 17. PMID 31694954
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-N-0145.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of HIV were recruited from the NIH Clinical Center and the local HIV community. Recruitment started on 4/1/2018 and ended on 11/22/2020.
Pre-assignment Details: 68 individuals were pre-screened and 13 individuals met the eligibility criteria and expressed interest in participating in the study.
Groups:
- HIV Participants: Participants who received 200mg Pembrolizumab administered as a one-time intravenous infusion.
Period: Overall Study
Arm/Group | HIV Participants
Started | 13
Completed | 6
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | HIV Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Grade 3 or Higher Adverse Events
Description: The frequency of Grade 3 and higher Adverse Events (AEs) that are probably or definately causal to pembrolizumab was calculated for the duration of the study, i.e., up to 52 weeks following infusion of pembrolizumab.
Time Frame: study duration (up to 52 weeks post infusion)
Measure: Number; unit: number of occurrences
Groups:
- HIV Participants: Participants who received 200 mg Pembrolizumab administered as a one-time intravenous infusion
Arm/Group | HIV Participants
Number analyzed (Participants) | 6
number of occurrences | 0

2. Secondary Outcome: Change in HIV-specific Antibody Responses in the CSF and Serum Using LIPS Assay.
Description: Analysis of the effects of pembrolizumab on various immunologic responses (antigens) was conducted at baseline and 3 weeks after infusion of pembrolizumab.
  Antibody responses have been correlated with cure responses in the "Berlin patient". Utilizing the "Berlin patient's" antibody levels as a benchmark for the post-treatment of the study participants, a change in the following antigens was analyzed at 3 weeks post-infusion of pembrolizumab, in CSF and serum: p24, Matrix, gp120, Reverse transcriptase, Integrate, Protease, and pg41. A positive value suggests exposure to the HIV protein; while a negative value suggests no exposure to the HIV protein.
Time Frame: 3 weeks after infusion
Measure: Mean (Standard Deviation); unit: Fold change
Groups:
- Serum Antibody Levels: Change in serum antibody levels at 3 weeks post-infusion compared to baseline
- CSF Antibody Levels: Change in CSF antibody levels at 3 weeks post infusion compared to baseline
Arm/Group | Serum Antibody Levels | CSF Antibody Levels
Number analyzed (Participants) | 6 | 6
Fold change
  p24 | 0.99 (0.15) | 1.32 (0.76)
  Matrix | 1.05 (0.20) | 0.87 (0.38)
  gp120 | 1.06 (0.31) | 1.13 (0.86)
  Reverse transcriptase | 0.95 (0.11) | 1.35 (1.06)
  Integrase | 0.99 (0.18) | 0.87 (0.50)
  Protease | 0.99 (0.23) | 1.29 (0.96)
  gp41 | 1.07 (0.15) | 0.95 (0.29)

3. Secondary Outcome: Change in CSF Cytokine Profile Post-study Drug
Description: A change in CSF cytokine profile was measured between baseline and 3 weeks after infusion of pembrolizumab. Cytokines are proteins that communicate with and trigger the immune system to attack invaders in the body. An increase in an individual cytokine level after 3 weeks suggests an immune reaction.
Time Frame: 3 weeks after infusion
Measure: Mean (Standard Deviation); unit: Fold change
Groups:
- HIV Participants: Participants who received 200 mg of Pembrolizumab administered as a one-time intravenous infusion.
Arm/Group | HIV Participants
Number analyzed (Participants) | 6
Fold change
  EGF | 1 (0)
  Eotaxin | 1.68 (1.34)
  G-CSF | 1 (0)
  GM-CSF | 1 (0)
  IFNa2 | 1 (0)
  IFNg | 1 (0)
  IL-10 | 1.42 (1.02)
  IL-12P40 | 1.49 (1.25)
  IL-12P70 | 1 (0)
  IL-13 | 1 (0)
  IL-15 | 0.92 (0.38)
  IL-17A | 1 (0)
  IL-1RA | 1.27 (0.67)
  IL-1a | 1.45 (1.31)
  IL-1b | 1 (0)
  IL-2 | 1 (0)
  IL-3 | 1 (0)
  IL-4 | 1 (0)
  IL-5 | 1 (0)
  IL-6 | 1 (0)
  IL-7 | 1 (0)
  IL-8 | 0.97 (0.26)
  IP-10 | 1.47 (1.11)
  MCP-1 | 2.05 (2.36)
  MIP-1a | 0.93 (0.26)
  MIP-1b | 1.16 (0.54)
  RANTES | 1 (0)
  TNFa | 1 (0)
  TNFb | 1 (0)
  VEGF | 1 (0)

4. Secondary Outcome: Peripheral CD4 Counts
Description: A change in peripheral CD4 counts was measured from baseline to 3 weeks post-infusion of pembrolizumab. CD4 T cells help coordinate the immune response by stimulating other immune cells, such as macrophages, B lymphocytes (B cells), and CD8 T lymphocytes (CD8 cells), to fight infection. HIV weakens the immune system by destroying CD4 cells. CD4 counts in the blood were measured at baseline and 3 weeks after infusion of pembrolizumab. A positive value suggests an increase in the CD4 count while a negative value suggests a decrease in the CD4 count.
Time Frame: 3 weeks after infusion
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | HIV Participants
Number analyzed (Participants) | 6
percent change | -66.33 (241.87)

5. Secondary Outcome: HIV RNA in Plasma and CSF
Description: Change in HIV RNA levels was measured in plasma and CSF from baseline to 3 weeks after pembrolizumab infusion. A positive change value suggests an increase in viral load, while a negative change value suggests a decrease in viral load.
Time Frame: 3 weeks after infusion
Population: Unable to verify the data from one participant, potentially skewing the results measuring the HIV RNA in CSF.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- HIV RNA Level in Serum: Change in CD4+ HIV RNA level in serum at baseline and week 3
- HIV RNA Level in CSF: Change in CD4+ HIV RNA in CSF at baseline and Week 3
Arm/Group | HIV RNA Level in Serum | HIV RNA Level in CSF
Number analyzed (Participants) | 6 | 5
percent change | 8.66 (9.3) | 16276.6 (36382.17)

6. Secondary Outcome: Change in FDG-PET/CT Metabolic Uptake in CNS
Description: Change in FDG-PET/CT metabolic uptake in the CNS from baseline to 3 weeks after infusion of pembrolizumab was measured. A change reflecting an increase in update might suggest higher metabolic activity in that brain region, while a change reflecting a decrease in uptake might suggest lower metabolic activity in that brain region.
Time Frame: 3 weeks after infusion
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | HIV Participants
Number analyzed (Participants) | 6
percent change
  Whole Brain | -0.85 (0.88)
  Caudate | -1.48 (1.88)
  Putamen | -1.28 (1.57)
  Thalamus | -1.14 (1.88)
  Frontal Lobe | -2.14 (1.98)

7. Secondary Outcome: Change in PD-1 Expression in the CSF and Blood Cells
Description: A change in PD-1 expression on CD4 and CD8 T cells in the CSF and blood cells, was measured from baseline to 3 weeks after infusion of Pembrolizumab. A decline in PD-1 expression on CD4 and CD8 T cells suggests more potential T cell targeting response.
Time Frame: 3 weeks after infusion
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- HIV Participants: Participants was received 200 mg of Pembrolizumab administered as a one-time intravenous infusion.
Arm/Group | HIV Participants
Number analyzed (Participants) | 6
percent change
  CD4+ in blood | -12.94 (5.42)
  CD8+ in blood | -4.06 (1.79)
  CD4+ in CSF | -14.05 (10.63)
  CD8+ in CSF | -9.99 (7.40)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the study duration beginning on day of infusion of Pembrolizumab up to week 52 post-infusion.
Description: Adverse events were collected during each study visit utilizing a study questionnaire, ensuring each participant was solicited in the same manner.
Groups:
- HIV Participants: Participants received 200mg Pembrolizumab administered as a one-time intravenous infusion.
Arm/Group | HIV Participants
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV Participants (N=6)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 3 (4)
Blood Bicarbonate Decreased (Investigations) | 2 (2)
Lipase Increased (Investigations) | 1 (1)
Cholesterol High (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03239899/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03239899/ICF_001.pdf